CLINICAL TRIAL: NCT06042881
Title: Retrospective Cohort Study of the Physiotherapy Procedure in Critically Ill Patients Diagnosed With COVID-19 During the First Wave
Brief Title: Retrospective Cohort Study of the Physiotherapy in Critically Ill Covid Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-COV-2022-36
Record Dates: First submitted 2023-08-07; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: physical therapy; covid; mechanical ventilation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective cohort study that will include patients from the ICU of the Hospital de la Santa Creu i Sant Pau in Barcelona during the period between March 11 and May 13, 2020. The cohorts are made up of two groups of patients admitted for severe COVID during the first wave, according to whether or not they received physiotherapy and the possible impact of physiotherapy on the days of mechanical ventilation in the two study groups will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COVID-19 in critical condition
* Adults >18 years
* Admission to the ICU from March 11 to May 13, 2020

Exclusion Criteria:

* Patients readmitted on 2 occasions during the study period, the second will be omitted income.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size obtained will not be from any formal calculation, it will be a sample per convenience of inclusion of all patients admitted to the ICU with a diagnosis of COVID-19 During the study period, 189 subjects, with whom it is expected to achieve the objectives of the study.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Days of mechanical ventilation | 2 months
  To evaluate the effectiveness of early physiotherapy in critically ill patients with COVID-19 admitted to the ICU in terms of reducing days of mechanical ventilation

SECONDARY OUTCOMES:
days of stay | 2 months
  Evaluate the days of stay in the ICU
Assess morbidity and mortality. | 2 months
  Assess morbidity and mortality.
Assess the comorbidities of patients admitted for COVID-19 in critical condition | 2 months
  Assess the comorbidities of patients admitted for COVID-19 in critical condition
PNS lesion in prono position | 2 months
  To know if there is a greater risk of suffering a PNS lesion the more rounds of pronation
Assess the comorbidities of patients admitted for COVID-19 in critical condition | 2 months
  To know if the delay in the prescription of physiotherapy (FST) influences the appearance of PNS lesions.
Start of standing in critrically ill | 2 months
  To evaluate the start of standing (BP) in critically ill patients infected with COVID-19 who underwent FST.
Workload in physiotherapy | 2 months
  To assess the workload of the cohort of patients who underwent physiotherapy during the first wave of COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain